CLINICAL TRIAL: NCT06420596
Title: A Randomised Controlled Trial on the Effectiveness of Remote App-assisted Physiotherapy in Patients With Non-specific Low Back Pain (RemotePT)
Brief Title: The Effectiveness of Remote App-assisted Physiotherapy in Patients With Non-specific Low Back Pain (RemotePT)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00430; mu24Netzer
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
Keywords: Physiotherapy; Remote app-assisted physiotherapy; Akina Cloud; Musculoskeletal assessment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control intervention (Other): In the control group, patients receive conventional physiotherapy.
  Interventions: Other: Conventional Physiotherapy
- Study Intervention (Experimental): In the interventional group, patients receive 12 weeks of a remote physiotherapy via Akina Cloud in addition to conventional physiotherapy (treatment according to FMH Switzerland guidelines). Patients are encouraged to complete at least three app-guided training sessions per week.
  Interventions: Other: Conventional Physiotherapy; Device: Akina Cloud

INTERVENTIONS:
Other: Conventional Physiotherapy — Conventional physiotherapy is one prescription of 9 in person physiotherapy sessions (according to FMH Switzerland guidelines). The frequency of the physiotherapy sessions are at the discretion of the treating clinician, but the recommendation is 1 to 2 sessions per week.
Device: Akina Cloud — Akina Cloud is a digital health application that supports therapeutic exercises in people with musculoskeletal disorders. It is the first app-supported physiotherapy solution available in Switzerland.
  Other Names: Remote physiotherapy
  Arms: Study Intervention

SUMMARY:
The aim of this single-center, observational randomised controlled trial is to evaluate the effectiveness of using Akina Cloud, a remote app-assisted physiotherapy, in managing non-specific low back pain among patients.

DETAILED DESCRIPTION:
In Switzerland, 1.5 million people suffer from low back pain (LBP), which is often the cause of disability. Non-specific LBP is a major cause of high healthcare costs in developed countries and often leads to early retirement.

The development of musculoskeletal assessment through remote app-assisted therapeutic home training may be useful for individuals with non-specific LBP, providing initial support for its implementation in primary care in the patient's home. App-supported therapeutic solutions allow healthcare professionals to prescribe and monitor rehabilitation programs remotely. These innovative solutions have the potential to reduce healthcare costs and provide clinical outcomes comparable or even better than conventional physiotherapy, especially for patients in remote areas.

Akina Cloud, a digital health application that supports therapeutic exercises in people with musculoskeletal disorders, is the first remote app-assisted therapeutic home training solution available in Switzerland. It provides patients with exercise and educational content and facilitates communication between patients and therapists via the application.

The aim of this single-center, observational randomised controlled trial is to show the efficacy of Akina Cloud-mediated physiotherapy in patients with non-specific LBP. Therefore, all enrolled patients receive one prescription of physiotherapy treatment, while patients in the intervention group in contrast to the control group additionally receive the Akina Cloud-mediated physiotherapy. The efficacy of the remote app-assisted physiotherapy through Akina Cloud in regards to reducing the functional disability (primary objective), reducing perceived pain and increasing quality of life (secondary objectives) in comparison to conventional physiotherapy alone is evaluated.

The results of the trial will demonstrate whether app-assisted therapeutic home training is promising approach for managing non-specific low back pain, with the potential to significantly impact patient outcomes and healthcare delivery in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of non-specific low back pain (International Classification of Diseases, 10th edition M54.5) with the pain duration of at least 6 weeks
* Low back pain score of >3 out of 0-10, based on the numerical pain rating scale at the time of enrolment
* Ability to provide informed consent and participation in the study
* Prescription for physiotherapy
* German speaking
* Presence of an email address, internet connection and a private laptop as well as being able to use the laptop

Exclusion Criteria:

* Inpatient pain therapy (red flags)
* History of lumbar spine surgery during the last year
* Known diagnosis of performance-limiting illnesses as psychological disorders, diseases of the cardiovascular system, etc.
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-06-19 (Estimated)

PRIMARY OUTCOMES:
Assessment of the functional disability | Baseline, 0.5, 4, 8, and 12 weeks
  The patient's functional disability is assessed using the Oswestry Disability Index (ODI). The ODI is a patient-completed questionnaire that provides a subjective percentage score indicating the level of disability in daily activities. Scores range from 0 to 100, with higher scores indicating greater disability. To evaluate whether the remote app-assisted physiotherapy using Akina Cloud in addition to conventional physiotherapy is more effective than conventional physiotherapy alone, the average ODI scores between the two groups are compared.

SECONDARY OUTCOMES:
Assessment of pain | Baseline, 0.5, 4, 8, and 12 weeks
  The pain intensity is assessed by asking the patient to rate his/her pain on a Numerical Rating Scale (ranging from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain). To evaluate whether the remote app-assisted physiotherapy using Akina Cloud in addition to conventional physiotherapy is more effective in reducing perceived pain than conventional physiotherapy alone, the average values between the two groups are compared.
Assessment of the quality of life by the Veterans RAND 12-Items Health Survey | 0.5, 4, 8, and 12 weeks
  The health-related quality of life is assessed using the Veterans RAND 12-Items Health Survey (VR-12), which measures various aspects of physical and mental health, generating Physical Component Summary and Mental Component Summary scores. Scores range from 0 to 100, with higher scores indicating better health outcomes. To evaluate whether the remote app-assisted physiotherapy using Akina Cloud in addition to conventional physiotherapy is more effective in increasing the quality of life than conventional physiotherapy alone, the average scores between the two groups are compared.

CONTACTS AND LOCATIONS:
Overall Officials: Cordula Netzer, PD Dr. med., Principal Investigator — Department of Spine Surgery, University Hospital Basel
Locations (1):
- Department of Spine Surgery, University Hospital Basel, Bethesda Spital, Basel, Canton of Basel-City, Switzerland